CLINICAL TRIAL: NCT01354184
Title: An International, Multi-centre, Randomised, Stratified, Double-blinded, Placebo-controlled, 4-parallel Group Trial Investigating the Efficacy and Safety of Three Different Dose Levels of CRD007 (The AORTA Trial)
Brief Title: CRD007 for the Treatment of Abdominal Aorta Aneurysm (The AORTA Trial)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RSPR Pharma AB (Industry)
Other Study IDs: Cardoz-003
Record Dates: First submitted 2011-05-13; First posted 2011-05-16 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

ARMS (4):
- CRD007 10 mg tablet (Experimental)
  Interventions: Drug: CRD007
- CRD007 25 mg tablet (Experimental)
  Interventions: Drug: CRD007
- CRD007 40 mg tablet (Experimental)
  Interventions: Drug: CRD007
- CRD007 matching placebo tablet (Placebo Comparator)
  Interventions: Drug: CRD007 matching placebo

INTERVENTIONS:
Drug: CRD007
  Arms: CRD007 10 mg tablet; CRD007 25 mg tablet; CRD007 40 mg tablet
Drug: CRD007 matching placebo
  Arms: CRD007 matching placebo tablet

SUMMARY:
This is an investigation of the efficacy and safety of CRD007 compared to placebo in the treatment of patients with abdominal aortic aneurysm.

ELIGIBILITY:
Inclusion Criteria:

* Infra-renal abdominal aortic aneurysm

Exclusion Criteria:

* Previous infra-renal aortic surgery
* Known diabetes

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Sillesen, MD DMSc, Principal Investigator — Rigshospitalet, Denmark
Locations (15):
- Denmark (5):
  - Aalborg Hospital, Department of Vascular Surgery V, Aalborg
  - Aarhus Universitetshospital Skejby, Hjerte-Lunge-Kar kir. afd. T, Aarhus
  - Rigshospitalet, Karkirurgisk afdeling RK 3111, Copenhagen
  - Sygehus Lillebælt, Karkirurgisk Forskningsenhed, Kolding
  - Regionshospitalet Viborg, Karkiurgisk Forskningssektion, Viborg
- Sweden (8):
  - Borås Hospital, Department of Surgery, Borås
  - Mälarsjukhuset, Team Kärl Kir. Klin., Eskilstuna
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Skånes Universitets Sjukhus, Institution of Surgical Science, Malmo
  - Universitetssjukhuset Örebro, Kirurgkliniken, Kärlsektionen, Örebro
  - Karolinska University Hospital, Kärlkirurgiska Kliniken, Stockholm
  - Uppsala University Hospital, Uppsala
  - Centrallaserettet, Kärlkirurgiska Kliniken, Västerås
- United Kingdom (2):
  - St George's Hospital NHS Trust, London
  - University Hospital of South Manchester, Manchester

REFERENCES:
- [Derived] Sillesen H, Eldrup N, Hultgren R, Lindeman J, Bredahl K, Thompson M, Wanhainen A, Wingren U, Swedenborg J; AORTA Trial Investigators. Randomized clinical trial of mast cell inhibition in patients with a medium-sized abdominal aortic aneurysm. Br J Surg. 2015 Jul;102(8):894-901. doi: 10.1002/bjs.9824. Epub 2015 May 12. PMID 25963302